CLINICAL TRIAL: NCT04849455
Title: Erector Spinae Plane Block Catheters: The Role in Acute Postoperative Pain After Hepatic Resection With Intrathecal Morphine
Brief Title: Erector Spinae Plane Block Catheters and Intrathecal Morphine for Hepatic Resection
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Engy T. Said, MD, Associate Clinical Professor, Anesthesiology., University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201661
Record Dates: First submitted 2021-03-25; First posted 2021-04-19 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Hepatic Resection; Acute Pain; Anesthesia; Anesthesia, Local
Keywords: acute postoperative pain; erector spinae plane block; liver resection
MeSH Terms: conditions — Acute Pain; Pain, Postoperative | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Active Treatment (Experimental): This group will receive a continuous erector spinae block catheter followed by an infusion of ropivacaine 0.2% at 10ml automatic set bolus per 120 minutes with 2ml/hr continuous infusion (14mls total every 2 hours per catheter)
  Interventions: Drug: 0.2% ropivacaine local anesthetic continuous erector spinae plane block; Drug: Spinal Morphine
- Placebo (Placebo Comparator): This group will receive a superficially placed (taped to the surface) erector spinae block catheter with a ropivacaine 0.2% infusion at 0.1ml /hr
  Interventions: Drug: 0.2% ropivacaine local anesthetic superficially taped continuous erector spinae plane block; Drug: Spinal Morphine

INTERVENTIONS:
Drug: 0.2% ropivacaine local anesthetic continuous erector spinae plane block — Treatment- continuous erector spinae block catheter followed by an infusion of ropivacaine 0.2% at 10ml automatic set bolus per 60 minute with 2ml/hr continuous infusion (12mls/hr total per catheter)
  Other Names: Treatment
  Arms: Active Treatment
Drug: 0.2% ropivacaine local anesthetic superficially taped continuous erector spinae plane block — Placebo- Superficially placed (taped to the surface) erector spinae block catheter with a ropivacaine 0.2% infusion at 0.1ml /hr
  Other Names: Placebo
  Arms: Placebo
Drug: Spinal Morphine — 200-300 mcg of spinal morphine

SUMMARY:
To determine whether the addition of erector spinae plane (ESP) catheters to existing multimodal analgesic regimen with intrathecal morphine provides superior postoperative analgesia in patients undergoing hepatic resection compared with patients not receiving ESP catheters.

DETAILED DESCRIPTION:
Hepatic resection surgery is especially painful and requires optimal postoperative pain control for early mobilization and improved respiratory function. While there are many options for pain control, including IV opioids and thoracic epidurals, their utility is often limited by decreased metabolism and coagulopathy respectively. Our institution's current regimen including multimodal analgesia combined with intrathecal morphine and physician discretion with ESP catheters to facilitate postoperative pain management. However, the duration of intrathecal morphine is 24 hours, which is not cover the duration of significant post-operative leading to an increase in intravenous opioid consumption. ESP block is a paraspinal fascial plane between the erector spinae muscle and the thoracic transverse processes blocking the dorsal and ventral rami of the spinal nerves. This provides a multi-dermatomal sensory block of the anterior, posterior and lateral thoracic and abdominal walls. The addition of a catheter allows for a continuous infusion of local anesthetic. In addition, unlike a hepatic resection with a thoracic epidural coagulation status is not a concern. We believe that if patients' have improved post-operative pain control they will have better participation in physical therapy, require less opioids and potentially have shorter hospital length of stay.

Specific Aim: To determine if the addition of ESP catheters to multimodal pain regimen with intrathecal morphine, would provide superior postoperative analgesia beyond the morphine's twenty-four hour duration in patients undergoing hepatic resection compared to patients not receiving ESP catheters.

Hypothesis 1: Patients undergoing hepatic resection will have improved postoperative analgesia - based on mean opioid consumption and numeric rating scale pain scores - during postoperative day (POD) 1, as defined by 24 hours after intrathecal morphine, to POD 3 following surgery when receiving routine multimodal analgesia with intrathecal morphine and multimodal pain management with addition of ESP catheters versus multimodal analgesia with intrathecal morphine alone.

Hypothesis 2: Patients undergoing hepatic resection will have decreased incidence of persistent postoperative pain - based on mean opioid consumption and standard of care numeric rating scale pain scores during their hospital stay and at home- when receiving routine multimodal analgesia with intrathecal morphine with addition ESP catheters versus multimodal analgesia with intrathecal morphine alone.

This will be randomized, subject-masked, placebo-controlled, human subjects clinical trial.

Enrollment. Consenting adults undergoing hepatic resection will be offered enrollment. Study inclusion will be proposed to eligible patients prior to surgery. If a patient desires study participation, written, informed consent will be obtained using a current UCSD Institutional Review Board (IRB)-approved Informed Consent Form (ICF). Selection for inclusion will not be based on gender, race, or socioeconomic status.

This will be a single-center (UCSD), randomized, controlled investigation.

Preoperative Procedures. Following written, informed consent, we will record baseline anthropomorphic information (age, sex, height, and weight) that is already provided by all patients having surgery. After consenting and prior to surgery, patients will be randomized (utilizing sealed envelopes with 1:1 ratio) to either intrathecal morphine and sham ESP catheters or intrathecal morphine and active ESP catheters. Currently the decision to place ESP catheters is at the discretion of the attending physician. The only difference for subjects participating in the study (vs those not participating) will be that the placement of ESP catheters and decision to activate them-currently standard-of-care and used daily at UCSD because of clinical equipoise-will be determined randomly, instead of the physician simply choosing him/herself.

Intrathecal morphine and sham ESP catheter group: In the preoperative holding area, all subjects in this cohort, will have a peripheral intravenous (IV) catheter inserted, standard noninvasive monitors applied, supplemental oxygen administered via a nasal cannula or face mask, and positioned sitting. Midazolam and fentanyl (IV) will be titrated for patient comfort, while ensuring that patients remain responsive to verbal cues. The area of insertion will be cleaned with iodine povacrylex and isopropyl alcohol (DuraPrep Surgical Prepping Solution, 3M St. Paul, MN USA), and a clear, sterile, fenestrated drape applied. After identifying with palpation the desired interspace using sterile techniques with the midline single shot spinal approach a 25g pencil point needle spinal needle is passed through an introducer needle. After free flow of cerebral spinal fluid (CSF) is established 300mcg of intrathecal morphine is slowly injected with additional aspiration of CSF at the midpoint and end of injection to confirm continued subarachnoid administration. Then bilateral T7-8 ESP catheters will be taped onto the patient's back after administration of local anesthetic at the site. The 0.2% ropivacaine infusions will be started at the ESP block catheter immediately after catheter insertion with a total rate of 0.1ml per hour.

Intrathecal morphine and ESP catheter group: Catheter insertion will adhere to current UCSD standard-of-care. In the preoperative holding area, all subjects in this cohort, will have a peripheral intravenous (IV) catheter inserted, standard noninvasive monitors applied, supplemental oxygen administered via a nasal cannula or face mask, and positioned sitting. In the preoperative holding area, all subjects in this cohort, will have a peripheral intravenous (IV) catheter inserted, standard noninvasive monitors applied, supplemental oxygen administered via a nasal cannula or face mask, and positioned sitting. Midazolam and fentanyl (IV) will be titrated for patient comfort, while ensuring that patients remain responsive to verbal cues. The area of insertion will be cleaned with iodine povacrylex and isopropyl alcohol (DuraPrep Surgical Prepping Solution, 3M St. Paul, MN USA), and a clear, sterile, fenestrated drape applied. After identifying with palpation the desired interspace using sterile techniques with the midline single shot spinal approach a 25g pencil point needle spinal needle is passed through an introducer needle. After free flow of CSF is established 300mcg (200mcg for age >65yrs or respiratory concerns) of intrathecal morphine is slowly injected with additional aspiration of CSF at the midpoint and end of injection to confirm continued subarachnoid administration. Then bilateral T7-8 ESP catheters will be placed under ultrasound guidance. A catheter will be placed with saline with 1:200,000 of epinephrine. To confirm catheter location 15 mls of 1% lidocaine with 1:200,000 epinephrine will be injected and the block sensory level will be confirmed with ice. A total of 30mls of 1% lidocaine with 1:200,000 epinephrine will be used for bilateral catheter placement (15mls per side). A Ropivacaine 0.2% infusions will be started at the ESP block catheter immediately after catheter insertion with a total rate of 12mls per hour, 2mls/hr continuous infusion and 10ml set bolus every 120mins.

Additional Postoperative Pain Interventions: Intraoperatively the patient will have general anesthesia. Postoperatively, both groups will be started on the same multimodal oral regimen and followed by the Acute Pain Service (APS) as per APS standard of care.

Current Standard Care: Currently, all patients undergoing hepatic resection receive preoperative intrathecal morphine and at the discretion of the attending anesthesiologist the patient may or may not receive ESP catheters as well as multimodal pain regimen managed by APS. Intraoperatively general anesthesia. The only difference for subjects participating in the study (vs those not participating) will be that they will be randomized to whether or not they get ESP catheters. We will ensure that there are no patient contraindications to either intervention.

Data collection: All data collection will be through standard UCSD nursing/therapy EPIC notes and patient interviews in-person during hospitalization or via telephone call.

ELIGIBILITY:
Inclusion Criteria:

* undergoing hepatic resection
* Admitting service requests APS consult
* >18 years old and able to provide consent

Exclusion criteria:

* pregnancy
* incarceration
* inability to communicate with the investigators and hospital staff
* severe hepatic disease
* chronic high-dose opioid use (defined as daily use for more than 4 weeks prior to surgery of at least the equivalent of 20 mg oxycodone);
* BMI > 40 kg/m2
* allergy to study medications (lidocaine, ropivacaine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-05-24 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Total opioid requirement postoperative day (POD) 1-3 | Total use from post-operative day (POD) 1, as defined by 24 hours after intrathecal morphine, to POD 3 (3 days from admission to recovery unit)
  Morphine Milligram Equivalents

SECONDARY OUTCOMES:
Total opioid requirement postoperative day (POD) 0-4 | Total use from hospital admission to POD 4 (4 days after admission to recovery unit)
  Morphine Milligram Equivalents
Pain Score at rest and with cough | Post-Operative Day 0, 1, 2, 3, 4, 14, 30
  Average pain score on the 10-point numeric rating scale (0 being no pain, 10 worst pain)
Discharge opioids and refills. | Typically within 14days of admission, then at 14 days, and at 30 days.
  Amount of opioids prescribed at discharge and amount taken/refills while at home
Nausea | Post-Operative Day 0, 1, 2, 3, 4
  Defined by number of antiemetics administered
Time to ambulation | Post-Operative Day 0, 1, 2, 3, 4
  Able to get out of bed with physical therapy
Time to oral intake | Post-Operative Day 0, 1, 2, 3, 4
  Diet advancement
Hospital Length Of Stay | Total number of days requiring hospitalization for surgical procedure. Up to 1 month.
  From admission to hospital for surgery to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Engy T Said, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Pietri L, Siniscalchi A, Reggiani A, Masetti M, Begliomini B, Gazzi M, Gerunda GE, Pasetto A. The use of intrathecal morphine for postoperative pain relief after liver resection: a comparison with epidural analgesia. Anesth Analg. 2006 Apr;102(4):1157-63. doi: 10.1213/01.ane.0000198567.85040.ce. PMID 16551916
- [Background] Nair S, McGuinness S, Masood F, Boylan JF, Conlon NP. Erector Spinae Plane Blocks in Major Hepatopancreaticobiliary Surgery: A Case Series. A A Pract. 2019 Nov 1;13(9):332-334. doi: 10.1213/XAA.0000000000001069. PMID 31361665